CLINICAL TRIAL: NCT02960204
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of Emricasan, an Oral Caspase Inhibitor, in Subjects With Non-Alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension
Brief Title: Emricasan, an Oral Caspase Inhibitor, in Subjects With NASH Cirrhosis and Severe Portal Hypertension
Acronym: ENCORE-PH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Histogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IDN-6556-41; NCT04806750 (obsolete NCT alias)
Record Dates: First submitted 2016-07-29; First posted 2016-11-09 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2021-12

CONDITIONS: Cirrhosis; Portal Hypertension; Non-alcoholic Steatohepatitis
Keywords: cirrhosis; Portal Hypertension; Non-alcoholic Steatohepatitis; Liver cirrhosis
MeSH Terms: conditions — Fibrosis; Hypertension, Portal; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Emricasan (5 mg) (Active Comparator): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (5 mg) twice a day.
  Interventions: Drug: Emricasan
- Emricasan (25 mg) (Active Comparator): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (25 mg) twice a day.
  Interventions: Drug: Emricasan
- Emricasan (50 mg) (Active Comparator): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (50 mg) twice a day.
  Interventions: Drug: Emricasan
- Matching Placebo (Placebo Comparator): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with a matching placebo twice a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emricasan
  Arms: Emricasan (25 mg); Emricasan (5 mg); Emricasan (50 mg)
Drug: Placebo
  Arms: Matching Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled trial involving subjects with NASH cirrhosis and severe portal hypertension (defined as HVPG ≥12 mmHg as determined by the central reader assigned to this study). Upon successful screening, subjects will be randomized to receive either emricasan 50 mg BID, 25 mg BID, or 5 mg BID or matching placebo BID.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years or older, able to provide written informed consent and able to understand and willing to comply with the requirements of the study.
* Cirrhosis due to NASH with exclusion of other causes of cirrhosis (e.g. chronic viral hepatitis, alcoholic liver disease, etc.)
* Compensated cirrhosis OR Decompensated cirrhosis with no more than 1 prior significant decompensating event
* Severe portal hypertension defined as HVPG ≥12 mmHg
* Subjects who are on NSBB, nitrates, diuretics, lactulose, rifaximin, or statins must be on a stable dose for at least 3 months prior to Day 1
* Willingness to utilize effective contraception (for both males and females of childbearing potential) from Screening to 4 weeks after the last dose of study drug

Exclusion Criteria:

* Evidence of severe decompensation
* Severe hepatic impairment defined as a Child-Pugh score ≥10
* ALT (alanine transaminase) > 3 times upper limit of normal (ULN) or AST (aspartate transaminase) >5 times ULN during screening
* Estimated creatinine clearance <30 mL/min
* Prior transjugular intrahepatic portosystemic shunt or other porto-systemic bypass procedure
* Known portal vein thrombosis
* Symptoms of biliary colic, e.g. due to symptomatic gallstones, within the last 6 months, unless resolved following cholecystectomy
* Current use of medications that are considered inhibitors of OATP1B1 and OATP1B3 transporters
* Alpha-fetoprotein >50 ng/mL
* History or presence of clinically concerning cardiac arrhythmias, or prolongation of screening (pre-treatment) QTcF interval of >500 msec
* History of or active malignancies, other than those successfully treated with curative intent and believed to be cured
* Prior liver transplant
* Change in diabetes medications or vitamin E within 3 months of screening
* Uncontrolled diabetes mellitus (HbA1c >9%) within 3 months of screening
* Significant systemic or major illness other than liver disease
* HIV infection
* Use of controlled substances (including inhaled or injected drugs) or non-prescribed use of prescription drugs within 1 year of screening
* If female: planned or known pregnancy, positive urine or serum pregnancy test, or lactating/breastfeeding
* Previous treatment with emricasan or active investigational medication (except methacetin) in a clinical trial within 3 months prior to Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2019-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette M Wetzel, Study Director — Histogen; Samuel Mboggo, Study Director — Histogen; Ruqayyah Abdulrahoof, Study Director — Histogen
Locations (30):
- United States (19):
  - Pasadena, Pasadena, California
  - Rialto, Rialto, California
  - Palmetto Bay, Palmetto Bay, Florida
  - Atlanta, Atlanta, Georgia
  - Clive, Clive, Iowa
  - Baltimore, Baltimore, Maryland
  - Detroit, Detroit, Michigan
  - Rochester, Rochester, Minnesota
  - Saint Paul, Saint Paul, Minnesota
  - Kansas City, Kansas City, Missouri
  - Durham, Durham, North Carolina
  - Philadelphia, Philadelphia, Pennsylvania
  - Germantown, Germantown, Tennessee
  - Arlington, Arlington, Texas
  - Houston, Houston, Texas
  - San Antonio, San Antonio, Texas
  - Norfolk, Norfolk, Virginia
  - Richmond, Richmond, Virginia
  - Seattle, Washington, Seattle, Washington
- Germany (5):
  - Bonn, Bonn
  - Halle (Saale), Halle
  - Leipzig, Leipzig
  - Mainz, Mainz
  - Münster, Münster
- Spain (6):
  - Barcelona, Barcelona
  - San Sebastian, Donostia / San Sebastian
  - Madrid, Madrid
  - Majadahonda, Majadahonda
  - Santander, Santander
  - Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share this data with outside researchers

REFERENCES:
- [Result] Garcia-Tsao G, Bosch J, Kayali Z, Harrison SA, Abdelmalek MF, Lawitz E, Satapathy SK, Ghabril M, Shiffman ML, Younes ZH, Thuluvath PJ, Berzigotti A, Albillos A, Robinson JM, Hagerty DT, Chan JL, Sanyal AJ; IDN-6556-14 Investigators(double dagger). Randomized placebo-controlled trial of emricasan for non-alcoholic steatohepatitis-related cirrhosis with severe portal hypertension. J Hepatol. 2020 May;72(5):885-895. doi: 10.1016/j.jhep.2019.12.010. Epub 2019 Dec 21. PMID 31870950

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants were excluded from the study and not randomized if they withdrew consent or did not meet inclusion/exclusion criteria.
Groups:
- Emricasan (5 mg): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (5 mg) twice a day.
  Emricasan
- Emricasan (25 mg): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (25 mg) twice a day.
  Emricasan
- Emricasan (50 mg): Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with emricasan (50 mg) twice a day.
  Emricasan
- Matching Placebo: Subjects with Non-alcoholic Steatohepatitis (NASH) Cirrhosis and Severe Portal Hypertension will be administered orally with a matching placebo twice a day.
  Placebo
Period: Overall Study
Arm/Group | Emricasan (5 mg) | Emricasan (25 mg) | Emricasan (50 mg) | Matching Placebo
Started | 65 | 65 | 66 | 67
Randomized | 65 | 65 | 66 | 67
Completed Week 24 of Study | 62 | 62 | 60 | 66
Completed Week 48 of Study | 55 | 55 | 50 | 59
Completed (Follow-Up) | 36 | 44 | 37 | 38
Not Completed | 29 | 21 | 29 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emricasan (5 mg) | Emricasan (25 mg) | Emricasan (50 mg) | Matching Placebo | Total
Number analyzed (Participants) | 65 | 65 | 66 | 67 | 263
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 39 | 41 | 44 | 171
  >=65 years | 18 | 26 | 25 | 23 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (8.77) | 62.0 (8.81) | 59.5 (9.48) | 61.4 (7.90) | 60.8 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 33 | 45 | 150
  Male | 28 | 30 | 33 | 22 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 11 | 12 | 18 | 60
  Not Hispanic or Latino | 42 | 50 | 52 | 47 | 191
  Unknown or Not Reported | 4 | 4 | 2 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 58 | 58 | 60 | 64 | 240
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 7 | 5 | 4 | 3 | 19
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 57 | 54 | 212
  Germany | 3 | 1 | 1 | 3 | 7
  Spain | 4 | 7 | 4 | 5 | 20
  France | 5 | 3 | 4 | 2 | 14
  Switzerland | 2 | 4 | 0 | 3 | 9
Hepatic Venous Pressure Gradient [Mean (Standard Deviation); unit: mmHg] | 16.88 (3.573) | 17.25 (3.300) | 16.91 (3.545) | 16.81 (3.724) | 16.96 (3.586)
Taking Non-Selective Beta Blockers at Baseline [Count of Participants; unit: Participants]
  No | 37 | 39 | 40 | 40 | 156
  Yes | 28 | 26 | 26 | 27 | 107
Cirrhosis Baseline Status [Count of Participants; unit: Participants]
  Compensated Cirrhosis | 49 | 49 | 48 | 55 | 201
  Decompensated Cirrhosis | 16 | 16 | 18 | 12 | 62
Varices [Count of Participants; unit: Participants]
  None | 19 | 14 | 19 | 19 | 71
  Present - Small | 21 | 27 | 25 | 34 | 107
  Present - Medium | 21 | 16 | 14 | 6 | 57
  Present - Large | 4 | 7 | 8 | 7 | 26
  Present - Not Specified | 0 | 1 | 0 | 1 | 2
Compensated Status with Varices [Count of Participants; unit: Participants] — Population: Two subjects (one in 25 mg emricasan arm and one in placebo arm) did not have data available.
  Participants
    number analyzed (Participants) | 65 | 64 | 66 | 66 | 261
    Compensated with none/small varices | 32 | 29 | 32 | 42 | 135
    Compensated with medium/large varices | 17 | 19 | 16 | 12 | 64
    Decompensated with none/small varices | 8 | 12 | 12 | 11 | 43
    Decompensated with medium/large varices | 8 | 4 | 6 | 1 | 19
Model for End-Stage Liver Disease (MELD) Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 6.0 to 40.0, and higher MELD scores indicate more severe disease.
  units on a scale | 9.17 (2.673) | 9.06 (2.200) | 9.24 (2.512) | 8.40 (2.511) | 8.97 (2.489)
MELD Classification (Median Cut) [Count of Participants; unit: Participants] — Scores range from 6.0 to 40.0, and higher MELD scores indicate more severe disease.
  Participants
    <= 8 | 33 | 31 | 30 | 44 | 138
    >= 9 | 32 | 34 | 36 | 23 | 125
MELD Component: Total Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 1.27 (0.514) | 1.31 (0.482) | 1.39 (0.725) | 1.20 (0.600) | 1.29 (0.696)
MELD Component: Serum Creatine [Mean (Standard Deviation); unit: mg/dL] | 1.02 (0.079) | 1.01 (0.053) | 1.04 (0.160) | 1.02 (0.086) | 1.02 (0.102)
MELD Component: International Normalized Ratio [Mean (Standard Deviation); unit: mg/dL] — Patients are assigned a score from 6 to 40. Worst score of 6 equates to 90% 3-month survival rate, while a best score of 40 equates to 7% 3-month survival rate.
  mg/dL | 1.18 (0.167) | 1.16 (0.167) | 1.16 (0.115) | 1.14 (0.113) | 1.16 (0.128)
Child-Pugh Score [Mean (Standard Deviation); unit: units on a scale] — Scores range from 5 to 15, and higher Child-Pugh scores indicate more severe disease.
  units on a scale | 5.5 (0.96) | 5.5 (0.69) | 5.6 (0.86) | 5.4 (0.75) | 5.5 (0.82)
Child-Pugh Classification [Count of Participants; unit: Participants] — Scores range from 5 to 15, and higher Child-Pugh scores indicate more severe disease. A = scores from 5 to 6; B = scores from 7 to 9; C = scores from 10 to 15. Population: Two subjects (one in the 5 mg emricasan arm and one in the 25 mg emricasan arm) did not have data available.
  Participants
    number analyzed (Participants) | 64 | 64 | 66 | 67 | 261
    A | 56 | 59 | 55 | 61 | 231
    B | 7 | 5 | 11 | 6 | 29
    C | 1 | 0 | 0 | 0 | 1
Child-Pugh Component: Total Bilirubin [Count of Participants; unit: Participants] — Each component of the Child-Pugh scale is scored from 1 to 3, with 3 being the most severe.
  Participants
    1 | 58 | 61 | 59 | 64 | 242
    2 | 5 | 3 | 4 | 2 | 14
    3 | 2 | 1 | 3 | 1 | 7
Child-Pugh Component: Total Albumin [Count of Participants; unit: Participants] — Each component of the Child-Pugh scale is scored from 1 to 3, with 3 being the most severe.
  Participants
    1 | 49 | 52 | 51 | 57 | 209
    2 | 15 | 13 | 14 | 10 | 52
    3 | 1 | 0 | 1 | 0 | 2
Child-Pugh Component: Ascites [Count of Participants; unit: Participants] — Each component of the Child-Pugh scale is scored from 1 to 3, with 3 being the most severe.
  Participants
    1 | 58 | 61 | 57 | 62 | 238
    2 | 7 | 4 | 9 | 5 | 25
    3 | 0 | 0 | 0 | 0 | 0
Child-Pugh Component Hepatic Encephalopathy [Count of Participants; unit: Participants] — Each component of the Child-Pugh scale is scored from 1 to 3, with 3 being the most severe.
  Participants
    1 | 63 | 65 | 66 | 67 | 261
    2 | 2 | 0 | 0 | 0 | 2
    3 | 0 | 0 | 0 | 0 | 0
Child-Pugh Component: Prothrombin Time (or International Normalized Ratio) [Count of Participants; unit: Participants] — Each component of the Child-Pugh scale is scored from 1 to 3, with 3 being the most severe. Population: One subject in the 5 mg emricasan arm did not have data available.
  Participants
    number analyzed (Participants) | 64 | 65 | 66 | 67 | 262
    1 | 63 | 65 | 66 | 67 | 261
    2 | 1 | 0 | 0 | 0 | 1
    3 | 0 | 0 | 0 | 0 | 0
Gallstones [Count of Participants; unit: Participants] | 30 | 28 | 31 | 27 | 116
Cholecystectomy [Count of Participants; unit: Participants] | 24 | 16 | 20 | 26 | 86

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hepatic Venous Pressure Gradient (HVPG)
Description: To assess the mean change from baseline to Week 24 in hepatic venous pressure gradient (HVPG)
Time Frame: Baseline to Week 24
Population: Full analysis set (Multiple Imputation)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Emricasan (5 mg) | Emricasan (25 mg) | Emricasan (50 mg) | Matching Placebo
Number analyzed (Participants) | 61 | 62 | 56 | 64
mmHg | -0.48 (3.356) | -0.81 (3.669) | -0.70 (3.400) | -0.18 (3.028)

2. Secondary Outcome: Improvement of HVPG Response Using a 20% Reduction From Baseline
Description: To assess subjects who have at least a 20 percent reduction from baseline in HVPG
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Emricasan (5 mg) | Emricasan (25 mg) | Emricasan (50 mg) | Matching Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 67
participants
  >= 20% reduction in HVPG: Yes | 8 | 14 | 10 | 9
  >= 20% Reduction in HVPG: No | 53 | 48 | 46 | 55
  Unknown | 4 | 3 | 10 | 3

3. Secondary Outcome: Caspase 3/7
Description: To assess whether number of Caspase 3/7 biomarkers is affected by emricasan as compared to placebo
Time Frame: Baseline to Week 24, Baseline to Week 48
Population: Full Analysis Set (Observed Cases)
Measure: Mean (Standard Deviation); unit: RLU
Arm/Group | Emricasan (5 mg) | Emricasan (25 mg) | Emricasan (50 mg) | Matching Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 67
RLU
  Week 24: number analyzed (Participants) | 59 | 60 | 59 | 66
  Week 24 | -0.01 (0.475) | -0.40 (0.597) | -0.46 (0.663) | -0.04 (0.339)
  Week 48: number analyzed (Participants) | 49 | 50 | 49 | 58
  Week 48 | 0.13 (0.541) | -0.18 (0.665) | -0.48 (0.564) | 0.05 (0.373)

4. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: To assess whether amount of non-specific (ALT) biomarkers are affected by emricasan compared to placebo
Time Frame: Baseline to Week 24 and Baseline to Week 48
Population: Full Analysis Set (Observed Cases)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Emricasan (5 mg) | Emricasan (25 mg) | Emricasan (50 mg) | Matching Placebo
Number analyzed (Participants) | 65 | 65 | 66 | 67
U/L
  Week 24: number analyzed (Participants) | 58 | 61 | 58 | 66
  Week 24 | -7.83 (10.650) | -8.06 (10.542) | -7.06 (12.010) | -1.69 (12.907)
  Week 48: number analyzed (Participants) | 50 | 51 | 49 | 57
  Week 48 | -6.54 (11.917) | -4.16 (9.850) | -5.34 (11.153) | -2.97 (12.457)

ADVERSE EVENTS:
Time Frame: First day of study treatment through the follow-up phase (Week 28 for participants who received treatment through Week 24 OR Week 50 for participants who received treatment through Week 48).
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Emricasan (5 mg) | Emricasan (25 mg) | Emricasan (50 mg) | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 1/65 | 2/65 | 1/66 | 0/67
Serious Adverse Events (participants affected / at risk) | 15/65 | 23/65 | 21/66 | 16/67
Other Adverse Events (participants affected / at risk) | 59/65 | 62/65 | 57/66 | 61/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emricasan (5 mg) (N=65) | Emricasan (25 mg) (N=65) | Emricasan (50 mg) (N=66) | Matching Placebo (N=67)
Gastrointestinal disorders (Gastrointestinal disorders) | 6 (6) | 6 (6) | 3 (3) | 2 (2) — Esophageal varices, ascites, gastric ulcer haemorrhage, haemorrhoidal haemorrhage, small intestinal obstruction, upper gastrointestinal haemorrhage.
Infections and infestations (Infections and infestations) | 4 (4) | 7 (7) | 7 (7) | 3 (3) — Pneumonia, bacterial pyelonephritis, bronchitis, cellulitis, cystitis, gastroenteritis rotavirus, viral gastroenteritis, influenza, necrotizing fasciitis, sepsis, urinary tract infection
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 1 (1) | 2 (2) — Hepatocellular carcinoma, breast cancer, colon cancer, prostate cancer, renal cancer
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) — Asthma, dyspnoea, epistaxis, hepatic hydrothorax, interstitial lung disease, pulmonary embolism
Renal disorders (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) — Acute kidney injury, nephrotic syndrome.
Cardiac disorders (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Acute myocardial infarct, congestive heart failure
Blood disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Anemia, Coombs positive haemolytic anaemia, splenic vein thrombosis
Multi-organ failure (General disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1) — Death, localized oedema, multi-organ failure, non-cardiac chest pain, oedema peripheral, pyrexia
Acute hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1) — Acute hepatic failure, biliary colic, chlecystitis, granulomatours liver disease.
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) — Dysarthria, Guillain-Barre Syndrome, Hepatic encephalopathy, Seizure, Subarachnoid haemorrhage.
Tibial fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 2 (2) — Procedural pain, spinal cord compression fracture, subdural haematoma, tibial fracture, post-operative urinary retention, wrist fracture.
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Coombs positive haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Oesophagael varices haemorrhage (Gastrointestinal disorders) | 4 | 5 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Death (General disorders) | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecytitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Granulomatous liver disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis rotovirus (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Necrotizing fasciitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 3 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypervolemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Hepatocellular cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 2 | 2 | 0 | 2
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Porto pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emricasan (5 mg) (N=65) | Emricasan (25 mg) (N=65) | Emricasan (50 mg) (N=66) | Matching Placebo (N=67)
Gastrointestinal disorders (Gastrointestinal disorders) | 31 (31) | 38 (38) | 33 (33) | 39 (39) — Abdominal pain, ascites, colitis, constipation, diarrhoea, intestinal diverticulum, dyspepsia, gastric ulcer, gastritis, GERD, haematemesis, nausea, oesophageal varices haemorrhage, vomiting
Pneumonia (Infections and infestations) | 33 (33) | 39 (39) | 32 (32) | 32 (32) — Acute sinusitis, bacteremia, bronchitis, cellulitis, influenza, kidney infection, gastroenteritis, nasopharyngitis, pneumonia, respiratory tract infection, sepsis, urinary tract infection.
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6) | 3 (3) | 4 (4) — Hepatocellular carcinoma, Hepatic neoplasm, Breast cancer, colon cancer, prostate cancer, renal cancer, squamous cell carcinoma.
Hepatic encephalopathy (Nervous system disorders) | 15 (15) | 19 (19) | 20 (20) | 22 (22) — Asterixis, Dysarthria, Guillain-Barre Syndrome, Headache, Hepatic encephalopathy, Migraine, neuralgia, paraesthesia.
Acute kidney injury (Renal and urinary disorders) | 10 (10) | 10 (10) | 10 (10) | 10 (10) — Acute kidney injury, Haemorrhagic cystitis, haematuria, nephrolithiasis.
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 7 | 10
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 7 | 2 | 5 | 7
Abdominal pain upper (Gastrointestinal disorders) | 4 | 7 | 8 | 3
Ascites (Gastrointestinal disorders) | 4 | 9 | 4 | 8
Constipation (Gastrointestinal disorders) | 3 | 4 | 1 | 6
Diarrhea (Gastrointestinal disorders) | 10 | 7 | 6 | 13
Nausea (Gastrointestinal disorders) | 6 | 9 | 8 | 11
Esophageal varices hemorrhage (Gastrointestinal disorders) | 4 | 5 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 4 | 3 | 4
Asthenia (General disorders) | 6 | 1 | 4 | 3
Fatigue (General disorders) | 3 | 6 | 6 | 6
Edema peripheral (General disorders) | 9 | 14 | 8 | 8
Pyrexia (General disorders) | 2 | 5 | 3 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 0 | 1 | 1 | 4
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 1 | 5
Bronchitis (Infections and infestations) | 6 | 2 | 7 | 3
Cellulitis (Infections and infestations) | 3 | 4 | 4 | 4
Influenza (Infections and infestations) | 2 | 6 | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 4 | 4 | 5
Pneumonia (Infections and infestations) | 5 | 0 | 3 | 1
Sinusitis (Infections and infestations) | 4 | 3 | 2 | 4
Upper respiratory infection (Infections and infestations) | 4 | 4 | 4 | 5
Urinary tract infection (Infections and infestations) | 9 | 11 | 6 | 10
Fall (Injury, poisoning and procedural complications) | 2 | 4 | 3 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 6 | 5 | 2
Dizziness (Nervous system disorders) | 4 | 2 | 4 | 6
Headache (Nervous system disorders) | 3 | 7 | 7 | 5
Hepatic encephalopathy (Nervous system disorders) | 5 | 5 | 5 | 12
Anxiety (Psychiatric disorders) | 5 | 1 | 0 | 3
Insomnia (Psychiatric disorders) | 6 | 3 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 5 | 2
Pruritus generalized (Skin and subcutaneous tissue disorders) | 6 | 1 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 4
Hypotension (Vascular disorders) | 0 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or discussion must be approved by the Sponsor prior to release.

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT02960204/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT02960204/SAP_001.pdf